CLINICAL TRIAL: NCT04637438
Title: Fecal Microbiota Transplantation in Postoperative Crohn's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Joint Authority for Päijät-Häme Social and Health Care (Other); Kuopio University Hospital (Other); Helsinki University Central Hospital (Other); Tampere University (Other)
Responsible Party: Principal Investigator, Elina Jokinen, Doctor of Medical Science, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R20041
Record Dates: First submitted 2020-10-21; First posted 2020-11-19 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Crohn Disease
Keywords: Fecal Microbiota Transplantation
MeSH Terms: conditions — Crohn Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplantation (Active Comparator)
  Interventions: Other: Fecal Microbiota Transplantation
- Plasebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — FMT via colonoscopy
  Arms: Fecal Microbiota Transplantation
Other: Placebo — Water infusion via colonoscopy
  Arms: Plasebo

SUMMARY:
This pilot study aims to detect possible trends or signals suggesting efficacy of FMT on prevention of delay of POR, to determine the safety of FMT in post operative CD, and asses if a full randomised controlled trial is feasible in this setting. With microbiota analysis we aim to assess if changes in gut microbiota are related to disease course of CD after operation.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Able to provide written consent
* Stricturing and/or fistulizing Crohn's disease needing ileocecal or ileal resection

Exclusion Criteria:

* Pregnancy
* Active infection, abscess or fistula at the time of the first colonoscopy
* Life expectancy <1 year
* Unable to provide written consent
* Use on antibiotics or probiotics at the time of first colonoscopy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in endoscopic Rutgeerts score between first and second colonoscopy | 1 year
  Rutgeerts endoscopic score ranges from i0 indicating remission to i4 indicating severe post-operative relapse. Cut off value > i1 will be used to compare number on patients in intervention group and in placebo group.

SECONDARY OUTCOMES:
Safety of FMT using FinFMT-Questionnaire | 3 months, 12 months, 5 years
  Unvalidated survey including 20 questions.
Clinical activity of Crohn's disease using Harwey-Bradshaw Index | 6 months, 12 months, 5 years
  Scores of less that 5 indicate that the patient's Crohn's disease is in remission while scores higher than 16 indicate severe disease activity.
  Median scores will be compared between intervention group and placebo group.
Histologic activity of Crohn's Disease using modified Global Histological Activity Score | 1 years, 5 years
  The GHAS consists of eight items assessing acute and chronic inflammatory changes, epithelial damage and the extent of inflammation (i.e. the proportion of biopsy specimens affected). Each of the eight items is scored, with the totals subsequently added together. Maximum number 14 indicates histological activity. The median GHAS score will be compared between intervention group and placebo group.
Change of microbiota in stool samples and in intestinal biopsies | 6 weeks,12 weeks, 48 weeks, 5 years
  The relative abundances of taxonomic units in cases versus controls and different time points will be compared at the level of phylum, class, genus, species and OTU. Alpha diversity measures will be determined from the original unfiltered dataset by counting observed taxa (OTU richness) and by Chao1, ACE, Shannon, Simpson and Fisher indices; diversity will be compared between time points.cases and controls. Beta diversity will be assessed by examining the results of principle component analysis using multiple distance methods, if appreciable difference between cases and controls or time points will be noted, formal testing of clustering will be performed. To simplify complex bacteriome profiles, we will also sort each sample into enterotypes based on the leading components of their bacteriomes; the enterotypes will be tested as a predictor of the case-control or disease status of cases.
Patient reported outcome | 12 weeks, 48 weeks,years 5
  IBD symptom index (IBD-SI) questionnaire. Minimum number of points 0 indicating remission, maximum number of points 15 indicating active disease or flare.
Change in inflammatory marker CRP mg/l | 6 weeks,12 weeks, 24 weeks, 48 weeks, 5 years
  Median in intervention group versus plasebo group
Need for hospitalization | Through study completion, an avarage of 1 year and 5 years
  Avarage number of days spent in hospital in intervention group vs. plasebo group
Need for treatment escalation | Through study completion, an avarage of 1 year and 5 years
  Number of patients needing treatment escalation from thiopurines to TNF alfa blockers in intervention group versus plasebo group
F-calpro microg/g | 6 weeks,12 weeks, 24 weeks, 48 weeks, 5 years
  Median in intervention group versus plasebo group
Hb mg/l | 6 weeks,12 weeks, 24 weeks, 48 weeks, 5 years
  Median in intervention group versus plasebo group

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No